CLINICAL TRIAL: NCT07023068
Title: Clinical Application of PD-L1 Targeted Imaging Agent ⁶⁸Ga-DPA in the Diagnosis of Lung Cancer
Brief Title: ⁶⁸Ga-DPA in the Lung Cancer Diagnosis
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-PDL1
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancers
Keywords: PD-L1; lung cancer; PET/CT
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-DPA PEWT/CT (Experimental)
  Interventions: Diagnostic Test: 68Ga-DPA PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-DPA PET/CT — Use 68Ga-DPA PET/CT in the diagnosis of lung cancer

SUMMARY:
In previous studies, we synthesized a PD-L1-targeted molecular probe, ⁶⁸Ga-DPA, and developed a ⁶⁸Ga-DPA injection for clinical research. Preliminary studies demonstrated its favorable safety profile and excellent imaging performance. Leveraging the established strengths of the Department of Nuclear Medicine at Peking Union Medical College Hospital, we now plan to conduct an exploratory PET/CT imaging study in lung cancer patients. This study aims to provide an in vivo, non-invasive, and visualizable technique for detecting PD-L1 expression levels and spatial distribution in tumors. It will further validate the clinical utility of this technology, offering critical diagnostic insights for initial assessment and treatment efficacy evaluation in PD-L1-positive tumor patients undergoing PD-L1-targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, regardless of gender.
* Patients clinically confirmed or suspected of lung cancer, with pathological specimens obtainable via biopsy or surgery within the recent 2 months.
* At least one measurable target lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Expected survival >3 months.

Exclusion Criteria:

* Severe hepatic or renal dysfunction (serum creatinine >3.0 mg/dL or any liver enzyme level ≥5× upper limit of normal).
* Women who are planning pregnancy, pregnant, or breastfeeding.
* Inability to lie supine for 30 minutes.
* Claustrophobia or other psychiatric disorders.
* Intolerance to any clinical procedures in the study.
* Other conditions deemed ineligible by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-28 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2027-09-28 (Estimated)

PRIMARY OUTCOMES:
SUV | 0-180 minutes post-injection
  measured by PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- 100730, Beijing, China

IPD SHARING:
Plan to Share IPD: No